CLINICAL TRIAL: NCT03043144
Title: TASTE ESRD: Taste And Smell TEsting in End Stage Renal Disease
Brief Title: Taste And Smell TEsting in End Stage Renal Disease
Acronym: TASTE ESRD
Status: Withdrawn | Type: Observational
Why Stopped: Investigator leaving the institution
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katherine Lynch, Instructor in Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2016P000152
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Kidney Failure, Chronic; Olfaction Disorders; Taste Disorders; Malnutrition
MeSH Terms: conditions — Kidney Failure, Chronic; Olfaction Disorders; Taste Disorders; Malnutrition | interventions — c-MYC-associated zinc finger protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End stage renal disease: Observational study, no intervention
  Interventions: Other: Worsening of olfaction from enrollment visit to 6 months; Other: Worsening of taste from enrollment visit to 6 months; Other: Serum Zinc; Other: Chronic rhinosinusitis; Other: Dialysis adequacy; Other: Decayed missing filled teeth index (DMFT)

INTERVENTIONS:
Other: Worsening of olfaction from enrollment visit to 6 months — Worsening of olfaction from enrollment visit to 6 months will be evaluated for association with the primary and secondary outcomes
Other: Worsening of taste from enrollment visit to 6 months — Worsening of taste from enrollment visit to 6 months will be evaluated for association with the primary and secondary outcomes
Other: Serum Zinc — Serum zinc will be evaluated for association with taste and/or smell impairment
Other: Chronic rhinosinusitis — Chronic rhinosinusitis will be evaluated for association with smell impairment
Other: Dialysis adequacy — Dialysis adequacy will be evaluated for association with taste and/or smell impairment
Other: Decayed missing filled teeth index (DMFT) — DMFT will be evaluated for association with taste impairment

SUMMARY:
Malnutrition is an important complication of advanced kidney disease and impairment in smell and taste may affect nutritional status. This study will examine the association between impairment in smell and taste and nutritional and functional markers among patients with end stage renal disease, as well as risk factors for smell and taste impairment.

DETAILED DESCRIPTION:
People with advanced chronic kidney disease (CKD) are at risk for malnutrition, which is associated with significantly increased mortality. Impairments in olfaction and taste are under-recognized and under-addressed symptoms that affect this population. Olfaction and taste influence appetite and nutritional status and represent a unique target for study and intervention. Small cross-sectional studies have shown a higher prevalence of olfactory (up to 56%) and taste disturbances (up to 35%) among patients with CKD compared with the general population, but little is known about longitudinal change in olfaction and taste in this population. Additionally, there is a lack of understanding about why these sensory disturbances more commonly occur in people with CKD, although there is speculation that uremia may contribute.

This information gained from this study will address these gaps in knowledge by studying longitudinal changes in olfaction and taste and their associations with concurrent and future nutritional and functional status. Additionally this study will attempt to identify potentially modifiable risk factors associated with olfactory and taste impairment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* End-stage renal disease requiring chronic dialysis

Exclusion Criteria:

* Known allergy to quinine
* Presence of a pacemaker or internal defibrillator
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (aged 18 or older) who have end-stage renal disease requiring chronic dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
change in lean body mass | from 6 months to 1 year
  lean body mass will be determined by dual-energy X-ray absorptiometry scan

SECONDARY OUTCOMES:
change in hand grip strength | from 6 months to 1 year
  measured by dynamometer
change in the physical function score | from 6 months to 1 year
  measured by Standard-Form 36 version 2

OTHER OUTCOMES:
change in serum albumin | from 6 months to 1 year
  change in serum albumin
change in dietary intake | from 6 months to 1 year
  measured by a food frequency questionnaire
change in anthropometric measures | from 6 months to 1 year
  triceps skinfold thickness, mid arm circumference, and weight
change in serum cholesterol | from 6 months to 1 year
  change in serum cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Lynch, MD, SM, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided